CLINICAL TRIAL: NCT02360020
Title: Performance of the XLIMUS Sirolimus-eluting Coronary Stent In Very Complex Lesions
Brief Title: The XLIMUS-DES in Very Complex Lesions
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Clinica Mediterranea (Other)
Responsible Party: Principal Investigator, Carlo Briguori, Chief of Invasive Cardiology, Clinica Mediterranea
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: NCTCM03
Record Dates: First submitted 2015-02-02; First posted 2015-02-10 (Estimated); Last update posted 2016-05-10 (Estimated); Status verified 2016-05

CONDITIONS: Coronary Atherosclerosis Due to Calcified Coronary Lesion; Chronic Total Occlusion of Coronary Artery
Keywords: coronary stent; outcome

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (1):
- XLimus patients (Experimental): participants must have symptomatic ischemic heart disease attributable to critical (that is, >70% visual estimate) stenotic lesions of native coronary arteries. Inclusion criteria are 1) chronic total occlusion (CTO), 2) severe calcification, and 3) severe tortuosity. CTO is defined as the presence of TIMI 0 flow within the occluded segment and angiographic or clinical evidence of an occlusion duration of ≥3 months. Calcification is defined severe when larger than 3x vessel diameter, and comprising the vessel wall totally in two perpendicular views. Tortuosity is defined severe when: one or more bends >= 90°, or three or more bends of 45-90° proximal to the diseased segment.
  Interventions: Device: XLimus

INTERVENTIONS:
Device: XLimus — Techniques attempted for facilitating stent delivery in such a complex lesions are: maximize guide catheter support, optimize predilatation of the stenosis, use of a stiffer guidewire. Specific tricks include: a) buddy-wire; anchoring balloon; GuideLiner catheter. In case of severe calcification, rotational atherectomy was electively performed with the Rotablator® system (Boston Scientific Corporation, Natick, MA, U.S.A.). Following stent implantation, postdilatation is performed in all instances with a non-compliant balloon

SUMMARY:
Stent delivery failure occurs in 4% of all percutaneous coronary interventions (PCI) and >90% of these failures are due to vessel tortuosity and/or calcification. The XLIMUS eluting coronary stent (CARDIONOVUM GmbH, Bonn, Germany) is a new type of endovascular prostheses characterised by better mechanical properties than traditional DES. This is a prospective, non-randomized, single-center pilot study, aiming to evaluate the performance of the XLIMUS DES in severely complex coronary lesions in real-world clinical practice.

DETAILED DESCRIPTION:
All consecutive patients who will undergo elective PCI in native coronary arteries at the Clinica Mediterranea (Naples, Italy) will be considered for eligility. Study participants wiil require to have symptomatic ischemic heart disease attributable to critical (that is, >70% visual estimate) stenotic lesions of native coronary arteries. Inclusion criteria in this pilot study are 1) chronic total occlusion (CTO), 2) severe target vessel calcification, and 3) severe target vessel tortuosity. CTO is defined as the presence of TIMI 0 flow within the occluded segment and angiographic or clinical evidence or high likelihood of an occlusion duration of ≥3 months. Calcification is defined severe when larger than 3x vessel diameter, and comprising the vessel wall totally in two perpendicular views. Tortuosity is defined severe when it satisfies the following criteria: one or more bends of 90° or more, or three or more bends of 45-90° proximal to the diseased segment.

200 patients will be enrolled into the study. Stents will be implanted according to current clinical practice. Techniques attempted for facilitating stent delivery in such a complex lesions are: maximize guide catheter support, optimize predilatation of the stenosis, use of a stiffer guidewire. Specific tricks include: a) buddy-wire; anchoring balloon; GuideLiner catheter. In case of severe calcification, rotational atherectomy will be electively performed with the Rotablator® system (Boston Scientific Corporation, Natick, MA, U.S.A.). Following stent implantation, postdilatation will be performed in all instances with a non-compliant balloon. All patients will receive aspirin 325 mg and clopidogrel (75 mg daily) before stent deployment, with a loading dose (600 mg of clopidogrel) given to patients not pretreated. All patients will receive 70 IU/Kg intra-arterial bolus of unfractionated heparin in order to achieve and activated clotting time >250 seconds. Glycoprotein IIb/IIIa inhibitors will be administered according to operator preference. Estimated glomerular filtration rate (eGFR) will be calculated by applying the Levey Modification of Diet in Renal Disease (MDRD) formula. Chronic kidney disease was defined as a eGFR <60 ml/min/1.73 m2 .

XLIMUS eluting-stent is made of cobalt chromium L 605 and the stent is available in a 6-, 8-, or 10-cell structure design (closed cell architecture). The struts thickness is 73µm. The 6-cell design is for stenting of coronary artery diameter of 2.25mm-2.50mm, 8-cell structure is used for stenting of 2.75-3.50 mm artery diameters, and the 10-cell is for larger artery diameter lesions (up to 5mm). The XLIMUS has an innovative hydrophilic-coated shaft and an extra-low tip profile (crossing profile = 0.90 mm) to access the most tortuous lesions. The highly biocompatible polylactid acid (PLLA) drug containing release matrix degrades smoothly and provides an optimal release kinetic profile. Within 30 days, about 70% of the anti-proliferative drug is distributed into the surrounding arterial tissue of the stent struts, ensuring a highly effective inhibition of smooth muscle cell migration and proliferation. Pharmacokinetic study result confirm sustained anti-proliferative drug efficacy up to 120 days.

The primary objective of the study is the assessment of the clinical performance of the XLILMUS DES, using the following criteria 1) device success, defined as the ability to insert the stent into the target lesion and the attainment of <20% residual stenosis (by visual estimate), 2) lesion success, defined as attainment of <20% residual stenosis of the target lesion using any percutaneous method, and 3) procedural success, defined as lesion success without any in-hospital and MACE.

ELIGIBILITY:
Inclusion Criteria:

* chronic total occlusion (CTO)
* severe calcification
* severe tortuosity

Exclusion Criteria:

• coronary artery lesions non satisfying the inclusion criteria

Ages: 18 Years to 90 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 200 (Actual)
Dates: Start 2014-08; Primary Completion 2015-12 (Actual); Study Completion 2016-05 (Actual)

PRIMARY OUTCOMES:
Stent Performance | up to 1 month
  The primary objective of the study was the assessment of the clinical performance of the XLIMUS DES, using the following criteria 1) device success, defined as the ability to insert the stent into the target lesion and the attainment of <20% residual stenosis (by visual estimate), 2) lesion success, defined as attainment of <20% residual stenosis of the target lesion using any percutaneous method, and 3) procedural success, defined as lesion success without any in-hospital Man 30-day MACE

SECONDARY OUTCOMES:
Inhospital, 30-day and 1-year MACE | 1 year
  Major adverse cardiac events included death of any cause, nonfatal myocardial infarction, and repeated revascularization by PCI or surgery occurring within 30-day and 1-year. Myocardial infarction was defined as the presence of pathological and new Q waves on an ECG or as an increase in creatine kinase-myocardial band level to >3 times the upper limit of normal (ULN). Periprocedural myocardial infarction was defined as an increase of troponin I ≥5 times ULN. Target lesion revascularization was defined as a clinically-driven repeat percutaneous coronary angioplasty or coronary artery bypass surgery. Stent thrombosis was defined according to the Academic Research Consortium definitions

CONTACTS AND LOCATIONS:
Overall Officials: Carlo Briguori, Md, PhD, Principal Investigator — Clinica Mediterranea
Locations (1):
- Clinica Mediterranea, Naples, Naples, Italy

IPD SHARING:
Plan to Share IPD: Yes
We plan to present and publish the results in an international journal of interventional cardiology

REFERENCES:
- [Background] Nikolsky E, Gruberg L, Pechersky S, Kapeliovich M, Grenadier E, Amikam S, Boulos M, Suleiman M, Markiewicz W, Beyar R. Stent deployment failure: reasons, implications, and short- and long-term outcomes. Catheter Cardiovasc Interv. 2003 Jul;59(3):324-8. doi: 10.1002/ccd.10543. PMID 12822150
- [Background] Feldman T. Tricks for overcoming difficult stent delivery. Catheter Cardiovasc Interv. 1999 Nov;48(3):285-6. doi: 10.1002/(sici)1522-726x(199911)48:33.0.co;2-3. No abstract available. PMID 10525229
- [Background] Fernandes V, Kaluza GL, Godlewski B, Li G, Raizner AE. Novel technique for stent delivery in tortuous coronary arteries: report of three cases. Catheter Cardiovasc Interv. 2002 Apr;55(4):485-90. doi: 10.1002/ccd.10139. PMID 11948896
- [Background] Ashikaga T, Sakurai K, Satoh Y. Tools & Techniques: stent delivery in distal lesions. EuroIntervention. 2010 Nov;6(5):660-1. doi: 10.4244/EIJV6I5A109. No abstract available. PMID 21044922
- [Background] Kumar S, Gorog DA, Secco GG, Di Mario C, Kukreja N. The GuideLiner "child" catheter for percutaneous coronary intervention - early clinical experience. J Invasive Cardiol. 2010 Oct;22(10):495-8. PMID 20944191
- [Background] Rieu R, Barragan P, Garitey V, Roquebert PO, Fuseri J, Commeau P, Sainsous J. Assessment of the trackability, flexibility, and conformability of coronary stents: a comparative analysis. Catheter Cardiovasc Interv. 2003 Aug;59(4):496-503. doi: 10.1002/ccd.10583. PMID 12891615
- [Background] Schmidt W, Lanzer P, Behrens P, Topoleski LD, Schmitz KP. A comparison of the mechanical performance characteristics of seven drug-eluting stent systems. Catheter Cardiovasc Interv. 2009 Feb 15;73(3):350-60. doi: 10.1002/ccd.21832. PMID 19085917
- [Background] Morice MC, Colombo A, Meier B, Serruys P, Tamburino C, Guagliumi G, Sousa E, Stoll HP; REALITY Trial Investigators. Sirolimus- vs paclitaxel-eluting stents in de novo coronary artery lesions: the REALITY trial: a randomized controlled trial. JAMA. 2006 Feb 22;295(8):895-904. doi: 10.1001/jama.295.8.895. PMID 16493102
- [Background] Lohavanichbutr K, Webb JG, Carere RG, Solankhi N, Jarochowski M, D'yachkova Y, Dodek A. Mechanisms, management, and outcome of failure of delivery of coronary stents. Am J Cardiol. 1999 Mar 1;83(5):779-81, A9. doi: 10.1016/s0002-9149(98)00990-4. PMID 10080438
- [Background] Cantor WJ, Lazzam C, Cohen EA, Bowman KA, Dolman S, Mackie K, Natarajan MK, Strauss BH. Failed coronary stent deployment. Am Heart J. 1998 Dec;136(6):1088-95. doi: 10.1016/s0002-8703(98)70168-1. PMID 9842025
- [Background] Mortier P, De Beule M, Segers P, Verdonck P, Verhegghe B. Virtual bench testing of new generation coronary stents. EuroIntervention. 2011 Jul;7(3):369-76. doi: 10.4244/EIJV7I3A62. PMID 21729840
- [Background] Gyongyosi M, Yang P, Khorsand A, Glogar D. Longitudinal straightening effect of stents is an additional predictor for major adverse cardiac events. Austrian Wiktor Stent Study Group and European Paragon Stent Investigators. J Am Coll Cardiol. 2000 May;35(6):1580-9. doi: 10.1016/s0735-1097(00)00570-2. PMID 10807464
- [Background] Briguori C, Visconti G, Focaccio A, Donahue M. Performance of the XLIMUS sirolimus-eluting coronary stent in very complex lesions. Minerva Cardioangiol. 2014 Feb;62(1):1-8. PMID 24500212